CLINICAL TRIAL: NCT04667533
Title: A Phase 1, Open-Label, Single Dose, Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Desidustat for Treatment of Anemia in Patients Receiving Chemotherapy
Brief Title: Desidustat in the Treatment of Chemotherapy Induced Anemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zydus Lifesciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DESI.20.001
Record Dates: First submitted 2020-11-09; First posted 2020-12-14 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2020-11

CONDITIONS: Anemia of Chronic Kidney Disease; Chemotherapy Effect
Keywords: Chemotherapy induced Anemia
MeSH Terms: interventions — desidustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Desidustat tablet (Experimental)
  Interventions: Drug: Desidustat

INTERVENTIONS:
Drug: Desidustat — A total of 24 participants will be enrolled.
  The study is divided into three cohorts as given below:
  1. Cohort I: Single-dose 100 mg
  2. Cohort II: Single-dose 150 mg
  3. Cohort III: Single-dose 200 mg

SUMMARY:
This is a Phase 1, Open-label, Single Dose, Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Desidustat for treatment of anemia in patients receiving chemotherapy.

DETAILED DESCRIPTION:
A total of up to approximately 24 patients will be enrolled to receive Desidustat in an open-label manner.

The study is divided into three cohorts as given below:

1. Cohort I: Single-dose 100 mg
2. Cohort II: Single-dose 150 mg
3. Cohort III: Single-dose 200 mg

Note:- After evaluation of PK data of 100 mg dose cohort, next cohort with higher dose will be decided. Maximum dose of Desidustat will not be exceeded than 200 mg.

First cohort will be given 100 mg single dose of Desidustat. On completion of safety and PK evaluation of first cohort,the next cohort with escalated single dose (150 mg) of Desidustat will be initiated. Similar way third cohort with 200 mg single dose will be initiated after safety evaluation of 150 mg cohort data.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of non-myeloid malignancy.
2. Ability to comprehend and willingness to sign a written ICF for the study.
3. Male and Female patients at least 18 years old at the time of signing the ICF.
4. Anemia caused by cancer treatment (chemotherapy) defined as Hb ≤11.0 g/dL at screening.
5. Subjects with eGFR >60 mL/min/1.73 meter sequre at screening.
6. Weight should be ≥50 kg.
7. Willingness to participate after informed consent.
8. Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception.
9. Ability to swallow and retain oral medication.

Exclusion Criteria:

1. Known hypersensitivity to Desidustat and excipients in the investigational drug product.
2. History or presence of significant alcoholism, smoking or drug of abuse within 30 days at the time of screening.
3. History of RBC transfusion <4 weeks prior enrollment.
4. History or presence of any clinically significant electrocardiogram abnormalities during screening.
5. Cardiovascular risks, such as myocardial infarction, stroke, heart failure or thromboembolic event (e.g., deep vein thrombosis (DVT) or pulmonary embolism) within previous 6 months of screening
6. Major illness and/or major surgery in the last 3 months.
7. Planned elective surgery during the study
8. Receiving or has received any investigational drug within the 30 days before receiving Desidustat.
9. Any participants with poor peripheral venous access.
10. A positive test result for Human Immunodeficiency Virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibody at screening visit.
11. Female patients with following criteria will not be recruited:

    * History of pregnancy or lactation in the past 3 months
    * Fertile female volunteers not protected against pregnancy by adequate long-term antifertility measures
    * History of less than 1 year of menopause and not using adequate long-term anti-fertility measures
    * Using hormone replacement therapy
    * Unable to give assurance for protection against pregnancy for 3 months after the participation in this trial
    * Positive serum β-hCG level at the screening visit
12. Abnormal baseline laboratory investigations as follows:

    * WBC count ≤ 3 x 103/uL
    * Platelets count ≤ 100 x 103/uL
    * Bilirubin ≥ 1.5 mg/dL
    * ALT and/or AST ≥ 2.5 times of the ULN.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2022-03-27 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
To evaluate Adverse event of Desidustat following a single oral dose of 100 or 150 or 200 mg in patients with chemotherapy induced anemia. | Change from Baseline to Day 7 and Day 30
  The Common Terminology Criteria for Adverse Event (CTCAE) (Version 4.03 or higher) system will be used for reporting and grading

SECONDARY OUTCOMES:
Change of hemoglobin measurement from baseline | Change from baseline to Day 7 and Day 30
  a single oral dose of 100 or 150 or 200 mg in patients with chemotherapy induced anemia.

OTHER OUTCOMES:
Maximum plasma concentration (Cmax) | Change from Baseline to 72 hours in blood
  a single oral dose of 100 or 150 or 200 mg in patients with chemotherapy induced anemia.
  To compute pharmacokinetics, blood PK samples will be collected at pre-dose (<-0.5 h) and then 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 10.0, 12.0, 24.0, 48.0 and 72.0 hour post the single dose administration.
  Patients will be discharged on Day 1 and provide Day 2 and Day 3 PK as an outpatient visit for PK draws.
Time to reach maximum plasma concentration (Tmax) | Change from Baseline to 72 hours in blood
  a single oral dose of 100 or 150 or 200 mg in patients with chemotherapy induced anemia.
  To compute pharmacokinetics, blood PK samples will be collected at pre-dose (<-0.5 h) and then 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 10.0, 12.0, 24.0, 48.0 and 72.0 hour post the single dose administration.
  Patients will be discharged on Day 1 and provide Day 2 and Day 3 PK as an outpatient visit for PK draws.
Area under the curve from the time of dosing to the last measurable concentration (AUC0-t) | Change from Baseline to 72 hours in blood
  a single oral dose of 100 or 150 or 200 mg in patients with chemotherapy induced anemia.
  To compute pharmacokinetics, blood PK samples will be collected at pre-dose (<-0.5 h) and then 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 10.0, 12.0, 24.0, 48.0 and 72.0 hour post the single dose administration.
  Patients will be discharged on Day 1 and provide Day 2 and Day 3 PK as an outpatient visit for PK draws.
Terminal half life (t1/2) | Change from Baseline to 72 hours in blood
  a single oral dose of 100 or 150 or 200 mg in patients with chemotherapy induced anemia.
  To compute pharmacokinetics, blood PK samples will be collected at pre-dose (<-0.5 h) and then 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 10.0, 12.0, 24.0, 48.0 and 72.0 hour post the single dose administration.
  Patients will be discharged on Day 1 and provide Day 2 and Day 3 PK as an outpatient visit for PK draws.
Elimination rate constant (λz) | Change from Baseline to 72 hours in blood
  a single oral dose of 100 or 150 or 200 mg in patients with chemotherapy induced anemia.
  To compute pharmacokinetics, blood PK samples will be collected at pre-dose (<-0.5 h) and then 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 10.0, 12.0, 24.0, 48.0 and 72.0 hour post the single dose administration.
  Patients will be discharged on Day 1 and provide Day 2 and Day 3 PK as an outpatient visit for PK draws.
Clearance (CL) | Change from Baseline to 72 hours in blood
  a single oral dose of 100 or 150 or 200 mg in patients with chemotherapy induced anemia.
  To compute pharmacokinetics, blood PK samples will be collected at pre-dose (<-0.5 h) and then 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 10.0, 12.0, 24.0, 48.0 and 72.0 hour post the single dose administration.
  Patients will be discharged on Day 1 and provide Day 2 and Day 3 PK as an outpatient visit for PK draws.
Volume of distribution (Vd) | Change from Baseline to 72 hours in blood
  a single oral dose of 100 or 150 or 200 mg in patients with chemotherapy induced anemia.
  To compute pharmacokinetics, blood PK samples will be collected at pre-dose (<-0.5 h) and then 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 10.0, 12.0, 24.0, 48.0 and 72.0 hour post the single dose administration.
  Patients will be discharged on Day 1 and provide Day 2 and Day 3 PK as an outpatient visit for PK draws.
Amount recovered in Urine | Change from baseline to 24 hours in urine
  Urine PK collection will occur relative to dosing of Desidustat at pre-dose (within 2 hours before dosing) and then at the proposed time points (0-6, 6-12 and 12-24 hr) for clearance. Desidustat and the drug metabolite in urine and additional assay may be required.
Percent recovered in urine | Change from baseline to 24 hours in urine
  Urine PK collection will occur relative to dosing of Desidustat at pre-dose (within 2 hours before dosing) and then at the proposed time points (0-6, 6-12 and 12-24 hr) for clearance. Desidustat and the drug metabolite in urine and additional assay may be required.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Deven Parmar, MD, Study Chair — Cadila Healthcare Ltd.
Locations (1):
- HCG Manavata Cancer Centre,, Nashik, Mahar Ashtra, India

IPD SHARING:
Plan to Share IPD: No